CLINICAL TRIAL: NCT01807364
Title: Evaluation of Cardiovascular Risk Profile in Adult Patients With Congenital Adrenal Hyperplasia Due to 21-hydroxylase Deficiency Diagnosed During Childhood
Brief Title: Cardiovascular Risk Profile in Patients With Congenital Adrenal Hyperplasia
Acronym: cardiohcs
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 10032; P091106 (Other: APHP)
Record Dates: First submitted 2012-11-16; First posted 2013-03-08 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital adrenal hyperplasia (CAH); Cardiovascular risk; Microvascular dysfunction
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Congenital adrenal hyperplasia: Patients > 18 yrs with classical or non classical CAH diagnosed during childhood
- controls: control patients

SUMMARY:
Treatment with glucocorticoids and mineralocorticoids has changed congenital adrenal hyperplasia (CAH) from a fatal to a chronic lifelong disease. Long-term treatment, in particular the chronic (over-)treatment with glucocorticoids, may have an adverse effect on the cardiovascular risk profile in adult CAH patients. The objective of this study was to evaluate the cardiovascular risk profile of adult CAH patients.

DETAILED DESCRIPTION:
Treatment with glucocorticoids and mineralocorticoids has changed congenital adrenal hyperplasia (CAH) from a fatal to a chronic lifelong disease. Long-term treatment, in particular the chronic (over-)treatment with glucocorticoids, may have an adverse effect on the cardiovascular risk profile in adult CAH patients. The objective of this study was to evaluate the cardiovascular risk profile of adult CAH patients.

DESIGN: Case control study Primary objective : detection of cardiovascular damage in patients with classical or non classical CAH diagnosed in childhood. The patients will be compared with age- and gender- and tobacco status- matched control.

Secondary objective Study of microvascular function Evaluation of cardiovascular risk factors Total cumulative (TCG) and total average (TAG) glucocorticoid doses will be calculated from pediatric and adult files and correlated to arterial macro- and microcirculatory dysfunction.

Primary outcome Ultrasound evaluation of intima-media thickness at common carotids, carotid bulbs and left ventricular function Secondary outcome Peripheral and central blood pressure Skin capillary density and pulse-wave velocity Glucose and insulin during an oral glucose tolerance test Circulating cardiovascular risk markers (hsCRP, adiponectin, Interleukin-6) Lipid profile Anthropometry, fat and lean mass measured by dual-energy X-ray absorptiometry Total cumulative dose of glucocorticoid Number of subjects : 90 patients/90 controls Inclusion criteria of CAH patients

* Patients > 18 yrs with classical or non classical CAH diagnosed during childhood
* Absence of known cardiovascular disease
* Absence of combined oral contraceptives during the previous month Inclusion criteria of controls
* Age under 18
* Absence of known cardiovascular disease
* Absence of combined oral contraceptives during the previous month

Duration of the inclusion period: 3 years

ELIGIBILITY:
Inclusion criteria : patients

* Patients > 18 yrs with classical or non classical CAH diagnosed during childhood
* Absence of known cardiovascular disease
* Absence of combined oral contraceptives during the previous month

Inclusion criteria : controls

* Age > 18 yrs
* Absence of known cardiovascular disease
* Absence of combined oral contraceptives during the previous month

Exclusion criteria :

* Blood donation during the previous 3 months
* Cardiovascular disease
* Treatment by combined oral contraceptives
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients > 18 yrs with classical or non classical CAH diagnosed during childhood and controls
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-05; Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Ultrasound evaluation of intima-media thickness | day 1
  Ultrasound evaluation of intima-media thickness at common carotids, carotid bulbs and left ventricular function

SECONDARY OUTCOMES:
Blood pressure | day 1
  Peripheral
Skin capillary density | day 1
Insulin during an oral glucose tolerance test | day 1
Circulating cardiovascular risk markers | day 1
  Interleukin-6
Lipid profile | day 1
Lean mass measured by dual-energy X-ray absorptiometry | day 1
Total cumulative dose of glucocorticoid will be calculated from pediatric and adult files | day 1
  Calculated from pediatric and adult files
Pulse-wave velocity | day 1
Glucose during an oral glucose tolerance test | day 1
Anthropometry measured by dual-energy X-ray absorptiometry | day 1
Fat measured by dual-energy X-ray absorptiometry | day 1
Blood pressure | day 1
  Central
Circulating cardiovascular risk markers | day 1
  hsCRP
Circulating cardiovascular risk markers | day 1
  adiponectin

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bachelot, MD, PhD, Principal Investigator — APHP
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No